CLINICAL TRIAL: NCT07025759
Title: Effects of Peripheral Magnetic Stimulation on Cortical Excitability in Healthy Individuals
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Parameters_pMS
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy Individuals
Keywords: Peripheral Magnetic Stimulation; Cortical Excitabilty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Peripheral magnetic stimulation (90% + 1 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (90% of RMT + 1 Hz)
- Peripheral magnetic stimulation (100% + 25 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (100% of RMT + 25 Hz)
- Peripheral magnetic stimulation (90% + 25 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (90% of RMT + 25 Hz)
- Peripheral magnetic stimulation (100% + 1 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (100% of RMT + 1 Hz)
- Peripheral magnetic stimulation (100% + 10 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (100% of RMT + 10 Hz)
- Peripheral magnetic stimulation (110% + 1 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (110% of RMT + 1Hz)
- Peripheral magnetic stimulation (110% + 10 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (110% of RMT + 10Hz)
- Peripheral magnetic stimulation (110% + 25 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (110% of RMT + 25Hz)
- Peripheral magnetic stimulation (90% + 10 Hz) (Active Comparator)
  Interventions: Device: Peripheral magnetic stimulation (90% of RMT + 10 Hz)

INTERVENTIONS:
Device: Peripheral magnetic stimulation (90% of RMT + 1 Hz) — Low-frequency stimulation (1 Hz) at 90% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Peripheral magnetic stimulation (90% + 1 Hz)
Device: Peripheral magnetic stimulation (90% of RMT + 10 Hz) — High-frequency stimulation (10 Hz) at 90% of resting motor threshold intensity, totaling 2400 pulses.
  Arms: Peripheral magnetic stimulation (90% + 10 Hz)
Device: Peripheral magnetic stimulation (90% of RMT + 25 Hz) — High-frequency stimulation (25 Hz) at 90% of resting muscle threshold intensity, with 2400 pulses.
  Arms: Peripheral magnetic stimulation (90% + 25 Hz)
Device: Peripheral magnetic stimulation (100% of RMT + 1 Hz) — Low-frequency (1 Hz), at resting motor threshold intensity (100%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (100% + 1 Hz)
Device: Peripheral magnetic stimulation (100% of RMT + 10 Hz) — High-frequency (10 Hz), at resting motor threshold intensity (100%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (100% + 10 Hz)
Device: Peripheral magnetic stimulation (100% of RMT + 25 Hz) — High-frequency (25 Hz), at resting motor threshold intensity (100%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (100% + 25 Hz)
Device: Peripheral magnetic stimulation (110% of RMT + 1Hz) — Low-frequency (1 Hz), above resting motor threshold intensity (110%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (110% + 1 Hz)
Device: Peripheral magnetic stimulation (110% of RMT + 10Hz) — High-frequency (10 Hz), above resting motor threshold intensity (110%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (110% + 10 Hz)
Device: Peripheral magnetic stimulation (110% of RMT + 25Hz) — High-frequency (25 Hz), above resting motor threshold intensity (110%) protocol delivering 2400 pulses.
  Arms: Peripheral magnetic stimulation (110% + 25 Hz)

SUMMARY:
This study investigates the immediate effects of different parameters (frequency, intensity, and pulse number) of peripheral magnetic stimulation (rPMS) on cortical excitability in healthy individuals. Using a randomized, double-blind crossover design, the research aims to identify optimal stimulation protocols for modulating neural activity. Outcomes include measurements of motor-evoked potentials (MEPs), intracortical inhibition (ICI), and facilitation (ICF). Findings may enhance non-invasive therapeutic strategies for neurological disorders.

DETAILED DESCRIPTION:
This clinical trial is a crossover trial comparing 9 single-session rPMS protocols over the extensor carpi radialis muscle, testing three frequencies (1Hz, 10Hz, 25Hz), intensities (90%, 100%, 110% of resting motor threshold) across sequential phases.

Participants: Healthy adults (18-40 years) undergo pre-/post-intervention assessments: cortical (MEPs, ICI/ICF) excitability.

Design: Crossover, double-blind.

Analysis: ANOVA or Friedman tests (SPSS v20.0; α=0.05).

Significance: Clarifies parameter-specific neuromodulatory effects, guiding future rehabilitation protocols for neurological conditions.

Ethics: Approved by Federal University of Pernambuco's ethics committee (Resolution 466/12). Data stored securely for 5 years.

ELIGIBILITY:
Inclusion criteria: Healthy adults aged 18-40 years, both sexes, right-handed (confirmed via Edinburgh Handedness Inventory), and for females, consistent use of contraceptive medication to mitigate hormonal influences on nervous system excitability.

Exclusion criteria: Pregnancy; history of seizures or epilepsy; metallic implants in the head, spine, face, or heart; diagnosed neurological or musculoskeletal conditions interfering with assessments or interventions; or use of substances altering nervous system excitability.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Cortical excitabilty | Baseline (T0), immediately post-stimulation (T1), 15 minutes (T2), and 30 minutes (T3) post-stimulation.
  Cortical excitability will be assessed through motor-evoked potentials (MEPs) elicited by single-pulse transcranial magnetic stimulation (TMS) over the primary motor cortex (M1), targeting the first dorsal interosseous (FDI) representation area. The hotspot will be determined as the site producing the largest MEP amplitude at the lowest intensity, with stimulation delivered at 100% of the resting motor threshold (RMT). Additionally, paired-pulse TMS protocols will evaluate intracortical inhibition (ICI) and facilitation (ICF) using conditioning stimuli at 80% RMT (3 ms interstimulus interval for ICI, 10 ms for ICF) and test stimuli at 120% RMT. MEP amplitudes will be recorded via surface electromyography (EMG) from the FDI muscle using bipolar electrode placement, with signals sampled at 20,000 Hz (bandpass 5-10,000 Hz) to capture corticospinal excitability changes across timepoints (baseline, post-intervention, and follow-ups).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No